CLINICAL TRIAL: NCT03669185
Title: Pentaerithrityltetranitrat (PETN) Zur Sekundärprophylaxe Der Intrauterinen Wachstumsretardierung
Brief Title: Pentaerithrityl Tetranitrate (PETN) for Secondary Prevention of Intrauterine Growth Restriction
Acronym: PETN
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jena University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ZKS_0021PETN
Record Dates: First submitted 2018-08-28; First posted 2018-09-13 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Fetal Growth Retardation; Pregnancy Related; Intrauterine Growth Restriction
Keywords: PETN
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebos (Placebo Comparator): Placebos, 2 times daily 1 tablet, intake max. 133 days
  Interventions: Drug: Placebos
- Pentalong (Active Comparator): Pentalong, 2 times daily 1 tablet, intake max. 133 days
  Interventions: Drug: Pentalong

INTERVENTIONS:
Drug: Pentalong — Pentalong, 2 x daily 1 tablet, intake max. 133 days
  Other Names: Pentaeritrithyl tetranitrate; Pentalong® 50 mg
  Arms: Pentalong
Drug: Placebos — Placebos, 2 x daily 1 tablet, intake max. 133 days
  Arms: Placebos

SUMMARY:
Approximately 10% of all pregnancies experience mal perfusion of the placenta resulting in fetal growth restriction (FGR) of the fetus. FGR is the most important cause of perinatal mortality and morbidity. Impaired placental function determined by insufficient transformation of the uterine arteries and mal-perfusion of the placenta is the leading cause of FGR. So far, there is no treatment option for pregnancies complicated by FGR and the clinical management is restricted to close monitoring, assessing for the optimal time point of delivery of the fetus threatened by intrauterine death. In a pilot study a risk reduction of 38% for the development of severe FGR and FGR or death could be demonstrated by giving the organic nitrate pentaerithrityl-tetranitrate (PETN) to patients recognized at risk for FGR by impaired uterine artery Doppler at mid gestation (Schleussner, 2014). To confirm these results this prospective randomized placebo controlled double-blinded multicentre trial, was initiated.

DETAILED DESCRIPTION:
Affecting approximately 10% of pregnancies, fetal growth restriction (FGR), is the most important cause of perinatal mortality and morbidity. Impaired placental function determined by insufficient transformation of the uterine arteries and mal-perfusion of the placenta is the leading cause of FGR. So far, there is no treatment option for pregnancy complicated by FGR and the clinical management is restricted to close monitoring, assessing for the optimal time point of delivering the fetus threatened by intrauterine death. In a prospective randomized controlled trial a risk reduction of 38% (relative risk RR=0.609, 95% CI 0.367 to 1.011) for the development of IUGR and IUGR or death (RR=0.615, 95% CI 0.378 to 1.000) could be demonstrated by delivering the organic nitrate pentaerithrityl-tetranitrate (PETN) to patients recognized at risk for FGR by impaired uterine artery Doppler at mid gestation (Schleussner, 2014). To confirm these results a prospective randomized placebo controlled double-blinded multicentre trial was now initiated.

Eligible patients are pregnant women at risk of developing FGR meeting the inclusion criteria: abnormal uterine artery Doppler ultrasound, defined by a mean PI exceeding 1.6, singleton pregnancy, informed consent and 19+0 to 22+6 weeks of gestation. The composite endpoint of severe FGR (< birth weight below the 3rd centile) and intrauterine or neonatal death was defined as primary efficacy endpoint. and perinatal death. Key secondary endpoints are development of FGR (defined by birth weight < 10th percentile), severe FGR (< birth weight below the 3rd centile), intrauterine or neonatal death, placental abruption and preterm birth.

ELIGIBILITY:
Inclusion Criteria:

* abnormal uterine artery Doppler at 19+0 to 22+6 weeks of gestation, defined by a mean pulsatility index (PI) Exceeding 1.6
* singleton pregnancy
* age>/= 18 years
* informed consent

Exclusion Criteria:

* known fetal chromosomal or suspected major structural defects at time of enrollment
* premature rupture of membranes at time of enrolment; maternal disease defined as contraindication for intake of PETN
* anamnestic known insensitivity to Pentalong® or its ingredients or to medications with similar chemical structure
* participation of the patient in another clinical trial (parallel or within the waiting period of a previous clinical trial)
* multiple pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women between pregnancy week 19+0 and 22+6
Enrollment: 324 (Estimated)
Dates: Start 2017-07-26 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants who develop intrauterine/fetal growth restriction or perinatal death. | 19 weeks of pregnancy - seventh day of life
  Efficiency of PETN to prevent the development of intrauterine/fetal growth restriction or perinatal death.

SECONDARY OUTCOMES:
severe morbidity | 19 weeks of pregnancy - seventh day of life
  severe morbidity as a combined result of severe FGR (birth weight below the 3rd or 5th percentile) or perinatal death or premature abruption of placenta
birth weight | 19-40 weeks of pregnancy
  percentage of children with birth weight below the 3rd, 5th or 10th percentile
Number of participants who developed FGR | 19-40 weeks of pregnancy
  Number of participants who developed FGR, which necessitates delivery before 30 and 34 week of gestation
admission to NICU | Birth to discharge from the hospital
  rate of newborns transferred to neonatal intensive care unit
infant outcome | birth to discharge from NICU
  rate of newborns with intraventricular cerebral haemorrhage (grade II - IV) or necrotizing enterocolitis, b.o.
number of premature deliveries | 19 to 37 weeks of gestation
  number of premature deliveries before completed 34 and 37 weeks of gestation
mortality | 19 weeks of pregnancy - seventh day of life
  number of perinatal deaths

CONTACTS AND LOCATIONS:
Overall Officials: Tanja Groten, PD Dr., Principal Investigator — Universital Hospital Jena
Locations (14):
- Germany (14):
  - Universitäts-Frauenklinik Tübingen, Tübingen, Baden-Wurttemberg
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Klinikum der Universität München, München, Bavaria
  - Städtisches Klinikum München, München, Bavaria
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Universitätsklinikum Dresden, Dresden, Saxony
  - Uniklinikum Leipzig, Leipzig, Saxony
  - Krankenhaus St. Elisabeth und St. Barbara, Halle, Saxony-Anhalt
  - Universitätsklinik Halle, Halle, Saxony-Anhalt
  - Universitätsklinikum Schleswig Holstein, Kiel, Schleswig-Holstein
  - Universitätsklinikum Jena, Jena, Thuringia
  - Berlin Charité Campus Mitte, Berlin
  - Berlin Vivantes Klinikum Neukölln, Berlin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Groten T, Lehmann T, Stadtler M, Komar M, Winkler JL, Condic M, Strizek B, Seeger S, Jager Y, Pecks U, Eckmann-Scholz C, Kagan KO, Hoopmann M, von Kaisenberg CS, Hertel B, Tauscher A, Schrey-Petersen S, Friebe-Hoffmann U, Lato K, Hubener C, Delius M, Verlohren S, Sroka D, Schlembach D, de Vries L, Kraft K, Seliger G, Schleussner E; PETN study group. Pentaerythrityl tetranitrate improves the outcome of children born to mothers with compromised uterine perfusion-12-months follow-up and safety data of the double-blind randomized PETN trial. Am J Obstet Gynecol MFM. 2024 Apr;6(4):101332. doi: 10.1016/j.ajogmf.2024.101332. Epub 2024 Mar 7. PMID 38460823
- [Derived] Groten T, Lehmann T, Schleussner E; PETN Study Group. Does Pentaerytrithyltetranitrate reduce fetal growth restriction in pregnancies complicated by uterine mal-perfusion? Study protocol of the PETN-study: a randomized controlled multicenter-trial. BMC Pregnancy Childbirth. 2019 Sep 14;19(1):336. doi: 10.1186/s12884-019-2456-7. PMID 31521118
- See also: PETN Website — https://www.uniklinikum-jena.de/geburtsmedizin/petn.html
- See also: Publication Study Protocol — https://europepmc.org/article/PMC/PMC6744635